CLINICAL TRIAL: NCT04135079
Title: Immune Profiling in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Mario Boccadoro (Other)
Responsible Party: Sponsor-Investigator, Mario Boccadoro, Principal Investigator, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Other Study IDs: IMMUNE-UNITO
Record Dates: First submitted 2019-07-04; First posted 2019-10-22 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: immune transcriptome profile; Drop-seq; immune signatures; CyTOF; cytokine profile
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study propose to investigate the immune repertoire of MM patients at the time of diagnosis vs. 1st vs. 2nd vs. 3rd relapse. This study will provide insights into the immune status of MM patients before and after disease transformation and help identify patients who will benefit from immunotherapy. It will also allow us to predict the efficacy of these immune-mediated strategies and their associated toxicity. By understanding the immune-microenvironment in MM patients during disease progression, the investigator will be able to better design immunotherapeutic strategies for maximal success.

DETAILED DESCRIPTION:
Background: Immunotherapy has emerged as a new therapeutic strategy for the treatment of multiple myeloma (MM). The current immune-based strategies include the FDA-approved monoclonal antibodies elotuzumab1 and daratumumab2 targeting SLAMF7 and CD38 respectively, as well as immune approaches undergoing active clinical investigations such as bispecific T-cell engager,3 antibody-drug conjugate4 and cellular therapies like chimeric antigen receptor T cells.5-7 All of these treatment strategies are currently being tested in relapsed and refractory MM. However, MM patients, particularly those in the later stage of the disease, often have an impaired immune system.8-13 Given their curative potential, the investigator believe that immunotherapies should be used up front when the patient's immune system is still capable of mounting a normal immune response. Here the investigator propose to investigate the immune repertoire of MM patients at the time of diagnosis vs. 1st vs. 2nd vs. 3rd relapse. This study will provide insights into the immune status of MM patients before and after disease transformation and help identify patients who will benefit from immunotherapy. It will also allow us to predict the efficacy of these immune-mediated strategies and their associated toxicity. By understanding the immune-microenvironment in MM patients during disease progression, the investigator will be able to better design immunotherapeutic strategies for maximal success.

Samples: Peripheral blood samples from 20 newly diagnosed, 20 relapsed and/or refractory MM patients and 10 healthy donors will be collected before therapy. An additional peripheral blood sample will be collected at relapse in patients experiencing an early relapse (within 12 months from the start of therapy).

The project will include both a retrospective collection and a prospective collection of samples. Samples will be used for the current study after informed consent from the patient. The samples will be processed by Ficoll Paque gradient to isolate peripheral blood mononuclear cells (PBMCs). Peripheral blood serum will be collected as well.

Enrollment time: 9 months

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed MM patients or
* refractory MM patients or
* healthy donors.

Esclusion criteria:

* not newly diagnosed MM patients or
* not refractory MM patients or
* no healthy donors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: newly diagnosed, and/or refractory MM patients and healthy donors
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Determine the immune transcriptome profile in the peripheral blood of MM patients at diagnosis and relapse by bulk and single cell RNAseq. | through study completion, an average of 2 years
  PBMC samples will be subjected to bulk and single cell RNA sequencing for a comprehensive analysis of their immune transcriptomes, including but not limited to the gene expression profiles of high-resolution subsets of B cell, T cell, NK cell and myeloid compartments.

SECONDARY OUTCOMES:
Determine the immune signatures in the peripheral blood of MM patients at diagnosis and relapse by time-of-flight mass cytometry (CyTOF). | through study completion, an average of 2 years
  PBMCs will be subjected to CyTOF14, 15 for detailed immune cell analysis. All the major immune cell compartments including subsets of B cells, T cells, NK cells and myeloid cells will be assessed for their potential prognostic relevance in disease progression.

OTHER OUTCOMES:
Evaluate the cytokine profile in the peripheral blood of MM patients at diagnosis and relapse by cytokine arrays. | through study completion, an average of 2 years
  Peripheral blood serum will be subjected to cytokine arrays16 to screen for biomarkers that may predict potential adverse effects such as a cytokine storm. This cytokine profiling can potentially be used as a predictor of therapy-induced immune response, and thereby a treatment response. The cytokines that will be assessed are: 4-1BB, 4-1BB ligand, APRIL, B7-1, B7-2, B7-H1, B7-H2, BAFF, BCMA, CD27, CD40, CD40L, Fas, Fas L, Ferritin, GM-CSF, HVEM, ICOS, IFNg, IL10, IL12p40, IL12p70, IL-15, IL-17, IL-1b, IL-2, IL-2 Ra, IL-2 Rg, IL-4, IL-5, IL-6, IL-7, IL-8, L-selectin, MIP-1a, PD-1, PECAM-1, TGFb1, TIM-3, TNFa

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Larocca, Principal Investigator — S.C. Ematologia U
Locations (1):
- Aou Citta' Della Salute E Della Scienza Di Torino, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: Undecided